CLINICAL TRIAL: NCT03088839
Title: Observational Case-Control Study to Identify Circulating miR-218 as a Possible Non-invasive Biomarker of Amyotrophic Lateral Sclerosis (ALS)
Brief Title: Circulating Biomarker for Amyotrophic Lateral Sclerosis (ALS)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Neuromed IRCCS (Other)
Responsible Party: Principal Investigator, Alba Di Pardo, Dr., Neuromed IRCCS
Other Study IDs: ADP_01
Record Dates: First submitted 2017-03-13; First posted 2017-03-23 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS)
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 30 ALS patients
- 30 healthy controls

SUMMARY:
Amyotrophic Lateral Sclerosis (ALS) is a rare disease with a worldwide incidence of 2-3 cases per 100,000 individuals/year and it is characterized by progressive neurodegeneration of motor neurons. When motor neurons degenerate the ability of the brain to initiate and control muscle movement is lost. ALS manifests in two forms: Familiar ALS (FALS) with inherited risk genotypes, accounts for only 10% of cases and sporadic ALS (SALS) without apparent heritability accounts for 90% of cases. ALS can occur in both female and male subjects at any age but is more common in people aged over 40.

Although the molecular mechanism underlying the pathogenesis of ALS is still under investigation, recent research has revealed that diseases affecting motor neurons may be associated to alterations of RNA metabolism and biogenesis of small non-coding micro RNAs (miRNAs). miRNAs are circulating molecules, whose expression profiles are widely described to have an important potential in monitoring the progression of a disease, to promote the development of more targeted therapies and/or to determine the effectiveness of treatments. Altered patterns of specific miRNAs expression have been described in several pathological conditions. Evidence shows a significant reduction in the levels of certain miRNAs also in patients with ALS. Among others, miRNA-218 has been described to play a critical role in the onset of motor neurons differentiation and in establishing cell identity and fate.

Changes in the levels of miRNA-218 in the serum of ALS patients may potentially provide useful tools to determine the possible association with this disease and to candidate it as indicator of disease progression.

ELIGIBILITY:
Inclusion Criteria:

* ALS patients admitted to Centre for Rare Diseases, IRCCS Neuromed,
* Patients diagnosed ALS within 6 months,
* Patients age between 20 years and 75 years old,
* Patients underwent to differential diagnosis using diagnostic tools (EMG, NCV, MRI) to exclude other diseases with similar signs and symptoms,
* Subjects able to communicate verbally or by using a non-verbal communication system.

Exclusion Criteria:

* Pregnant women,
* Subjects with malignant tumor,
* Subjects/Patients with others neurological or psychiatric disorders,
* Subjects/Patients with systemic diseases,
* Subjects/Patients with positive blood test for hepatitis B or C, or HIV,
* Patients included in other clinical trials,
* Subjects/Patients showing inability to understand the informed consent and the study's purpose

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 60 individuals (30 subjects clinically diagnosed as ALS patients and 30 healthy controls) will be recruited at Centre for Rare Diseases, IRCCS Neuromed
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Identification of circulating miR-218 as biomarker for ALS | 8 months
  Quantitative assessment of potential changes in the levels of miR-218 in the serum of ALS patients vs healthy controls

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Neuromed, Pozzilli, Italy

IPD SHARING:
Plan to Share IPD: No